CLINICAL TRIAL: NCT04818372
Title: A Phase I, Multiple Center, Open-label, Dose Escalation and Dose Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of CM313 in Subjects With Relapsed or Refractory Multiple Myeloma and Lymphoma
Brief Title: Dose Escalation and Expansion Study of CM313 in Subjects With Relapsed or Refractory Multiple Myeloma and Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CM313MM001
Record Dates: First submitted 2021-03-24; First posted 2021-03-26 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Multiple Myeloma; Lymphoma
MeSH Terms: conditions — Multiple Myeloma; Lymphoma | interventions — Dexamethasone; Lenalidomide

STUDY DESIGN:
Intervention Model Description: Dose Escalation: Modified 3+3 dose escalation design: an accelerated dose titration design followed by traditional 3+3 dose escalation design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose escalation (Experimental): Subjects enrolled in this arm will receive a single dose of CM313 followed by a 3-week period for DLT observation. After that subjects will have 6 infusions at weekly intervals.
  Dose escalation will be carried out according to a modified 3+3 dose-escalation design. Accelerated dose titration design will be used for the first 4 dose levels (0.006mg/kg, 0.06mg/kg, 0.3mg/kg and 1.0mg/kg) and then traditional 3+3 dose escalation design will be used for the following levels (2.0mg/kg, 4.0mg/kg, 8.0mg/kg, 16mg/kg and 24mg/kg).
  Interventions: Drug: CM313-Dose escalation
- Dose expansion _Cohort 1 (Experimental): This cohort will comprise subjects with RRMM. Subjects will receive the CM313 in combination with dexamethasone.
  Interventions: Drug: CM313; Drug: Dexamethasone
- Dose expansion _Cohort 2 (Experimental): This cohort will comprise subjects with RRMM and NDMM. Subjects will receive the CM313 in combination with Rd regimen.
  Interventions: Drug: CM313; Drug: Dexamethasone; Drug: Lenalidomide

INTERVENTIONS:
Drug: CM313-Dose escalation — Subjects will receive a single dose of CM313 followed by a 3-week period for DLT observation. After that subjects will have 6 infusions at weekly intervals.
  Arms: Dose escalation
Drug: CM313 — Subjects will have 8 infusions at weekly intervals, and then 8 infusions at bi-weekly intervals. After that CM313 will be given every 4 weeks until disease progression or unacceptable toxicity.
  Arms: Dose expansion _Cohort 1; Dose expansion _Cohort 2
Drug: Dexamethasone — dexamethasone 40 mg/day at day 1,8,15,22 at 28 days cycle
  Arms: Dose expansion _Cohort 1; Dose expansion _Cohort 2
Drug: Lenalidomide — 25 mg/day lenalidomide 21 of 28 days cycle
  Arms: Dose expansion _Cohort 2

SUMMARY:
This is a multi-center, open-label, dose escalation and dose expansion, Phase 1 study to evaluate the safety, tolerability, PK and preliminary anti-tumor activity of CM313.

The dose escalation part will determine the MTD of CM313 in subjects with relapsed and/or refractory multiple myeloma (RRMM) or lymphoma based on a modified 3+3 dose escalation design (an accelerated dose titration design followed by traditional 3+3 dose escalation design).

The dose expansion part includes two cohorts. Cohort 1 will evaluate the safety and preliminary anti-tumor activity of CM313 in combination with Dexamethasone in subjects with RRMM. Cohort 2 will evaluate the safety and preliminary anti-tumor activity of CM313 in combination with Rd regimen (Lenalidomide/Dexamethasone) in subjects with RRMM or newly diagnosed MM (NDMM).

ELIGIBILITY:
Key Inclusion Criteria:

* Dose escalation: subjects with RRMM who have progressed on, or could not tolerate, all available established therapies and subjects with recurrent and refractory lymphoma.
* Dose expansion_cohort 1: subjects with RRMM who have progressed on, or could not tolerate, all available established therapies.
* Dose expansion_cohort 2: subjects with RRMM who have progressed on, or could not tolerate, all available established therapies, or subjects with NDMM.
* For MM: Documented initial diagnosis of multiple myeloma according to International Myeloma Working Group (IMWG) diagnostic criteria.
* For MM: Serum monoclonal paraprotein (M-protein) level greater than or equal to (>=) 0.5 gram per deciliter (g/dL) or urine M-protein level >=200 milligram per 24 hours (mg/24 h) or light chain multiple myeloma without measurable disease in the serum or the urine: serum immunoglobulin free light chain (FLC) >= 10 mg/dL and abnormal serum immunoglobulin kappa lambda FLC ratio.
* Eastern Cooperative Oncology Group (ECOG) performance status score <＝2.
* Women of childbearing potential and male subjects must agree to remain abstinent or use contraceptive methods as defined by the protocol.
* Side effects of any prior therapy or procedures for any medical condition has recovered to NCI-CTCAE v.5.0 Grade ≤ 1.

Key Exclusion Criteria:

* Previous treatment with any anti-CD38 therapy.
* Subjects with concurrent plasma cell leukemia.
* Received a cumulative dose of corticosteroids equivalent to greater than or equal to ( >=) 140 milligram (mg) of prednisone within the 14-day period before the first dose of study drug (does not include pretreatment medication).
* Vaccinated with live, attenuated vaccine within 4 weeks prior to the first dose.
* Received an allogenic stem cell transplant or an autologous stem cell transplant within 3 months before first dose of study drug.
* Central nervous system (CNS) involvement.
* The forced expiratory volume in one second (FEV1)<60%.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2021-04-26 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Dose escalation: Number of Participants with a Dose-Limiting Toxicity (DLT) | Up to 21 days after the first dose
Dose escalation and Dose expansion: Incidence, severity, and outcome of treatment emergent adverse events (TEAEs) and serious adverse events (SAEs) based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0 | Up to 30 days after the last dose of CM313 or until the start of subsequent anticancer therapy, if earlier
Dose expansion: To evaluate the activity of CM313 in combination with Rd/Dexamethasone as assessed by overall response rate (ORR) in RRMM patients | Up to 24 months
  ORR is defined as the proportion of participants who have a partial response (PR) or better according to the international myeloma working group (IMWG) criteria.

SECONDARY OUTCOMES:
Dose escalation: AUC to the last quantifiable concentration [AUC(0-last)], over the dosing interval [AUC(0-tau)], extrapolated to infinity [AUC(0-inf), time to Cmax (tmax), apparent half-life (t1/2), systemic clearance (CL). | 21 days after the first dose
Dose escalation and Dose expansion: AUC(0-last), AUC(0-tau), Cmax, t1/2, systemic clearance (CL), volume of distribution (Vz, Vss), minimum concentration (Cmin), Ctrough, accumulation ratios for Cmax and AUC(0-tau) for multiple doses | up to 24 months
Dose escalation and Dose expansion: Incidence of anti-CM313 | up to 24 months
Dose escalation: Overall Response Rate (ORR) | up to 24 months
  ORR is defined as the proportion of participants who have a partial response (PR) or better according to the IMWG criteria.
Dose escalation and Dose expansion: Clinical Benefit Rate (CBR) | up to 24 months
  CBR is defined as the proportion of participants who have a minimal response (MR) or better according to the IMWG criteria.
Dose escalation and Dose expansion: Duration of Response (DOR) | From the date of initial documentation of a response to the date of first documented evidence of progressive disease (PD) (up to 24 months)
  DOR is defined as time from date of initial documentation of a response (PR or better) to date of first documented evidence of PD, per IMWG criteria.or better according to the IMWG criteria.
Dose escalation and Dose expansion: Time to Response (TTR) | From the date of initial documentation of a response to the date of first documented evidence of progressive disease (PD) (up to 24 months)
  TTR is defined as the time between date of first dose of study drug and the first efficacy evaluation that the participant has met all criteria for PR or better.
Dose escalation and Dose expansion: Progression-Free Survival (PFS) | up to 24 months
  PFS is defined as time from date of first dose of study drug to date of first documented PD, per IMWG criteria, or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Wenming Chen, Dr., Principal Investigator — Beijing Chao Yang Hospital
Locations (3):
- China (3):
  - Beijing Chao-Yang Hospital, Capital Medical University (West Branch), Beijing, Beijing Municipality
  - Beijing Chao-Yang Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No